CLINICAL TRIAL: NCT03275480
Title: Institut Paoli Calmettes Myelodysplastic Syndromes Database
Status: Recruiting | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: BDD-SMD-IPC
Record Dates: First submitted 2017-09-06; First posted 2017-09-07 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Database of Institut Paoli-Calmettes patients diagnosed with Myelodysplastic Syndromes

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of Myelodysplastic Syndromes

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with new diagnosis of Myelodysplastic Syndromes
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-01-18 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Survival of patients with myelodysplastic syndrome(MDS) | 10 years
  Overall survival of all patients with MDS who are taken in charge in Institut Paoli Calmettes Cancer Center

SECONDARY OUTCOMES:
Collection of patients characteristics | 10 years
  Collection of characteristics of patients treated at Institut Paoli Calmettes in order to set up prospective and retrospective studies

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Vey, Pr, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, PACA, France